CLINICAL TRIAL: NCT01761071
Title: Time Serial Analysis on Preemptive Analgesia of Preoperative Topical Diclofenac and Ketorolac in Photorefractive Keratectomy(PRK)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 4-2012-0440
Record Dates: First submitted 2012-12-31; First posted 2013-01-04 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Myopes Who Have Undergone PRK.
MeSH Terms: interventions — Ketorolac; Ketorolac Tromethamine; Diclofenac; lactitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- group KO (Experimental): (ketorolac 0.5% in one eye, ofloxacin 0.3% in the other eye)
  Interventions: Drug: topical ketorolac 0.5% (Acular®, Allergan Inc, Irvine, CA)
- group DO (Active Comparator): (diclofenac 0.1% in one eye, ofloxacin 0.3% in the other eye)
  Interventions: Drug: topical diclofenac 0.1% (Voltaren®, Novartis, Bern, Switzerland)

INTERVENTIONS:
Drug: topical ketorolac 0.5% (Acular®, Allergan Inc, Irvine, CA) — On operation day, the patients were randomly assigned to one of the following two groups: group KO,preoperative application of topical ketorolac 0.5% (Acular®, Allergan Inc, Irvine, CA) in one eye and topical ofloxacin 0.3% (Ocuflox®, SamilInc, Seoul, Korea)in the other eye; group DO, topical diclofenac 0.1% (Voltaren®, Novartis, Bern, Switzerland) in one eye and ofloxacin 0.3% in the other eye. Neither the surgeon nor the participants knew which ophthalmic would go to which eye. A randomly assigned ophthalmic was instilled into right eye first three times by 1 minute interval 30 minutes prior to operation and the other ophthalmic was instilled into left eye with the same manner 10 minute later.
  Arms: group KO
Drug: topical diclofenac 0.1% (Voltaren®, Novartis, Bern, Switzerland) — On operation day, the patients were randomly assigned to one of the following two groups: group KO,preoperative application of topical ketorolac 0.5% (Acular®, Allergan Inc, Irvine, CA) in one eye and topical ofloxacin 0.3% (Ocuflox®, SamilInc, Seoul, Korea)in the other eye; group DO, topical diclofenac 0.1% (Voltaren®, Novartis, Bern, Switzerland) in one eye and ofloxacin 0.3% in the other eye. Neither the surgeon nor the participants knew which ophthalmic would go to which eye. A randomly assigned ophthalmic was instilled into right eye first three times by 1 minute interval 30 minutes prior to operation and the other ophthalmic was instilled into left eye with the same manner 10 minute later.
  Arms: group DO

SUMMARY:
The investigators performed this study to investigate pain prevention of preoperative topical nonsteroidal anti-inflammatory drug (NSAID) in photorefractive keratectomy(PRK) using time serial pain scoring.

ELIGIBILITY:
Inclusion Criteria:

1. at least 19 years of age
2. simultaneous bilateral PRK schedule
3. more than 400μm(including epithelium) of postoperative corneal thickness
4. less than 150μm of ablation depth.

Exclusion Criteria:

1. a history of ocular surgery or trauma
2. two-diopter more difference in spherical equivalent (SE) between the eyes, 3. keratoconus or other corneal pathology

4. use of systemic or topical NSAID within 1 month before the surgery 5. history of allergic reaction to aspirin or other NSAIDs 6. glaucoma or ocular hypertension (> 20 mmHg) 7. collagen vascular diseases 8. diabetic retinopathy 9. pregnancy or lactation 10. intraoperative complications.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2012-01; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Pain score using visual analog scale(VAS) of each topical NSAIDs pre-treated eyes. | Change the VAS level at 6, 18, 24, 36, 48, 72, and 96 hours after ketorolac in photorefractive keratectomy(PRK)
  Through these postoperative pain score which rated time serially, the effect of pre-treated topical NSAIDs(ketorolac and diclofenac) could be investigated on relieving postoperative pain after PRK.

CONTACTS AND LOCATIONS:
Locations (1):
- Departement of Ophthalmology, Yonsei University College of Medicine, Seoul, Seoul, South Korea